CLINICAL TRIAL: NCT03858283
Title: Mindfulness Based Health Care (MBHC) Program for Caregivers in the Neuropsychiatric Disorders in Alzheimer Patients and Anxiety and Depression in Caregivers
Brief Title: Mindfulness for Alzheimer Caregivers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the COVID pandemic, the lockdown in Spain began on 14 March 2020 and after two years we continue with contagion prevention measures that have not made it possible to implement face-to-face mindfulness courses or to evaluate participants.
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, ALICIA SANCHEZ PEREZ, Principal Investigator. Director of the Master's Degree in Occupational Therapy in Neurology, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mind01UMH
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Alzheimer Disease; Neurodegenerative Diseases; Dementia
Keywords: Mindfulness; Anxiety and depression symptoms; Caregivers; Alzheimer; neuropsychiatric disorders
MeSH Terms: conditions — Alzheimer Disease; Neurodegenerative Diseases; Dementia; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Health Care Program (Experimental)
  Interventions: Behavioral: Mindfulness Based Health Care (MBHC) Program
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness Based Health Care (MBHC) Program — Mindfulness Based Health Care (MBHC) Program for Caregivers of Alzheimer's Disease Patients. The duration of this group was 8 weeks. The program included one session per week, with each session lasting 1 hour and 30 minutes
  Arms: Mindfulness Based Health Care Program

SUMMARY:
Mindfulness Based Health Care (MBHC) includes meditation techniques to help caregivers of Alzheimer patients to be made more aware of their experience in the present moment. Half of the caregivers will learn the practice of mindfulness meditation once a week through 8 classes, and the other half will not receive any therapy. The primary purpose of this study is to explore the effects of this mindfulness program for caregivers on the neuropsychiatric symptoms in Alzheimer patients, as well as on anxiety and depression symptoms in their caregivers. Secondarily, to examine the effect of this program on cognitive function, daily activity living and quality of life in Alzheimer patients, as well as on the burden of caregiving, quality of life, psychological well-being, occupational balance, executive function and self-compassion in their caregivers.

DETAILED DESCRIPTION:
Alzheimer's disease is a progressive brain disorder that involves the loss of the ability to live independently, functional capacity and safety. Thus, patients often suffer neuropsychiatric disorders and need help from another person to live every day. Due to the burden of caregiving, the main caregivers can have anxiety and depression symptoms. With this scenario, we will conduct this randomized controlled trial aimed to evaluate the effect of mindfulness program for caregiver's vs control group on: 1) neuropsychiatric disorders, cognitive function, daily activity living and quality of life in Alzheimer patients; 2) anxiety and depression symptoms, burden of caregiving, quality of life, psychological well-being, occupational balance, executive function and self-compassion in their caregivers.

ELIGIBILITY:
Inclusion Criteria of Caregivers:

* be a caregiver of Alzheimer disease patient
* age over 18 years
* Score Mini Mental State Examination ≥26 points

Inclusion Criteria of Patients:

* Score of Scale Global Deterioration from 3 to 7 points (inclusive)
* Alzheimer disease diagnostic
* Non-institutionalized

Exclusion Criteria:

* Patient or caregivers with central nervous system disease with a neurological alteration (acquired brain damage, epilepsy, traumatic brain injury, multiple sclerosis and other movement disorders).
* Patient or caregivers with current or past history of alcohol or drug abuse
* Patient or caregivers with visual or hearing impairment
* Patient or caregivers with serious psychiatric illness (depression, psychosis, schizophrenia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Changes in Neuropsychiatric disorders of Alzheimer patients measured with Neuropsychiatric inventory | baseline, 8 weeks, 3 months after the 8 weeks
  Neuropsychiatric inventory includes 12 neuropsychiatric symptom domains: delusions, hallucinations, agitation/aggression, dysphoria/depression, anxiety, euphoria/elation, apathy/indifference, disinhibition, irritability/lability, aberrant motor behaviors, nighttime behavioral disturbances, and appetite/eating disturbances. Neuropsychiatric manifestations within a domain are collectively rated by the caregiver in terms of both frequency (1 to 4) and severity (1 to 3), yielding a composite symptom domain score (frequency×severity). Frequency and severity rating scales have defined anchor points to enhance the reliability of caregiver responses. Caregiver distress is rated for each positive neuropsychiatric symptom domain on a scale anchored by scores of 0 (not distressing at all) and 5 (extremely distressing).
Changes in Anxiety and depression symptoms in Caregivers of Alzheimer patients measured with Hospital Anxiety and Depression scale | baseline, 8 weeks, 3 months after the 8 weeks
  The Hospital Anxiety and Depression includes 14 items assessing anxiety (7-item) and depression (7-item), which are rated on a 4-point Likert-type (from 0 to 3). The scores in each subscale are computed by summing the corresponding items, with maximum scores of 21 for each subscale. A score of 0-7 is considered as normal, 8-10 as a borderline case, and 11-21 as a case (anxiety or depression)

SECONDARY OUTCOMES:
Changes in Cognitive Function of Alzheimer patients with Mini Mental State Examination | baseline, 8 weeks, 3 months after the 8 weeks
  The Mini Mental State Examination is composed of 13 items to assess with scores (0,1,2,3,4,5) according answer. the main objective is to briefly assess the mental state and allow observe the degree of progression of cognitive status through the following areas: orientation, fixation, concentration and calculation, memory, language and construction.
Changes in Executive Function of Alzheimer patients with Frontal Assessment Battery | baseline, 8 weeks, 3 months after the 8 weeks
  The FAB consists of 6 subtests that explore each of the processes controlled by the frontal lobes: 1) similarities (abstract reasoning/conceptualization); 2) lexical fluency (mental flexibility [i.e. self-organization, strategy and change]); 3) motor series (programming and motor planning); 4) conflicting instructions (sensitivity to interference); 5) Go-no-go test (inhibitory control and impulsiveness); and 6) prehension behavior (ability to inhibit a response to sensorial stimulation [i.e. environmental autonomy]). Higher scores of the test imply a better performance, and the total maximum score that can be obtained in the FAB is 18. The scoring is calculated by adding up the points for each test, which ranges from 0 to 3
Changes in Functional Capacity of Alzheimer patients with Disability Assessment for Dementia | baseline, 8 weeks, 3 months after the 8 weeks
  The Disability Assessment for Dementia is composed by 40 items that assess 4 basic ADLs (BADL: hygiene, dressing, continence, and eating; 17 items), and 6 instrumental activities (preparing of meals, use of telephone, finance and correspondence, medication, and leisure and domestic activities; 23 items). The items also reflect cognitive dimensions of functional capacity in terms of executive functioning: Initiative (13 items), planning and organization (10 items), and execution (17 items)
Changes in Quality of Life of Alzheimer patients with Quality of Life in Alzheimer's Disease scale | baseline, 8 weeks, 3 months after the 8 weeks
  The Quality of Life in Alzheimer's Disease scale uses 13 items a scale of 1-4 (poor, fair, good, or excellent) to rate a variety of life domains, including the patient's physical health, mood, relationships, activities, and ability to complete tasks. Total score range 13-52; higher scores indicate better Quality of life.
Change in Caregiver Burden of Caregivers of Alzheimer patients measured with Zarit Burden Interview | baseline, 8 weeks, 3 months after the 8 weeks
  Zarit Burden Interview consists of 22 items scored in 5-point Likert scale from 0 (never) to 4 (nearly always), except for the final item on global burden, rated from 0 (not at all) to 4 (extremely). The total score ranges from 0 to 88 with higher scores indicating higher burden.
Change in Occupational Balance of Caregivers of Alzheimer patients measured with Occupational Balance Questionnaire. | baseline, 8 weeks, 3 months after the 8 weeks
  Occupational Balance Questionnaire consists of 13 items scored in 6-point Likert scale from 0 (completely disagree) to 5 (completely agree). The total score ranges from 0 to 65 with higher scores higher occupational balance.
Change in Executive Function of Caregivers of Alzheimer patients measured with Frontal Assessment Battery | baseline, 8 weeks, 3 months after the 8 weeks
  The FAB consists of 6 subtests that explore each of the processes controlled by the frontal lobes: 1) similarities (abstract reasoning/conceptualization); 2) lexical fluency (mental flexibility [i.e. self-organization, strategy and change]); 3) motor series (programming and motor planning); 4) conflicting instructions (sensitivity to interference); 5) Go-no-go test (inhibitory control and impulsiveness); and 6) prehension behavior (ability to inhibit a response to sensorial stimulation [i.e. environmental autonomy]). Higher scores of the test imply a better performance, and the total maximum score that can be obtained in the FAB is 18. The scoring is calculated by adding up the points for each test, which ranges from 0 to 3
Change in Quality of Life of Caregivers of Alzheimer patients measured with Study Questionnaire Short Form 36 Health Survey | baseline, 8 weeks, 3 months after the 8 weeks
  The Study Questionnaire Short Form 36 Health Survey has eight scaled scores; the scoresare weighted sums of the questions in eachsection. Scores range from 0 -100 where lower scores =more disability and higher scores= less disability. This questionnaire include the follow subdimension: Vitality; Physical functioning; Bodily pain; General health perceptions; Physical role functioning; Emotional role functioning; Social role functioning; Mental health
Change in self-compassion of Caregivers of Alzheimer patients measured with Self-Compassion Scale | baseline, 8 weeks, 3 months after the 8 weeks
  Self-Compassion Scale measures the three components of self-compassion: shared humanity (SCSCH), mindfulness (SCS-M) and self-kindness (SCS-SK). It consists of 26 items evaluated with a Likert-type scale from 1 to 5 (1=almost never; 5=almost always). The total score is obtained with the sum of all items and ranges from 26 to 130 points.
Change in well-being of Caregivers of Alzheimer patients measured with Ryff's Well-being Scale | baseline, 8 weeks, 3 months after the 8 weeks
  Ryff's Well-being Scale measures psychological well-being. It is composed of 39 items that assess 6 dimensions: self-acceptance, autonomy, positive relationships with other people, personal growth, mastery of the environment, and purpose in life. The response format is a Likert-type scale from 1 (strongly disagree) to 6 (strongly agree). The range of the total score is 39 to 234 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Alicia Sánchez Pérez, Sant Joan d'Alacant, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided